CLINICAL TRIAL: NCT06806618
Title: Survey Evaluating the Burden and Management of HAE Crises by Patients and Caregivers
Brief Title: HAE Burden and Crisis Management
Acronym: ECRINS
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 3824.0394
Record Dates: First submitted 2025-01-28; First posted 2025-02-04 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Angioedema (HAE)
Keywords: survey; on-demand treatment; hereditary angioedema; burden; caregivers; quality of life
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with HAE: Patients will complete an online survey.

SUMMARY:
The study has been designed as a French, multicentric survey study to obtain data to describe the burden of on-demand treatment for patients with hereditary angioedema (HAE). The online survey assesses various aspects of HAE and in particular the burden of HAE from the patients' and caregivers' perspectives.

DETAILED DESCRIPTION:
The study has been designed as a French, multicentric survey study to obtain data to describe the burden of on-demand treatment for patients with hereditary angioedema (HAE). The study will also explore the burden related to the administration of intravenous or subcutaneous on-demand treatments. The study was designed to collect data concerning the burden of HAE in patients with HAE (during HAE attacks and between attacks) and in caregivers. The online survey will collect data to describe the characteristics of patients with HAE, the disease characteristics, details concern various aspects of HAE attacks, and the burden of HAE in patients and their caregivers.

ELIGIBILITY:
Inclusion Criteria:

For the patient population:

1. Patients with a confirmed diagnosis of HAE with a deficit in the C1 inhibitor.
2. Aged ≥12 years
3. Having consulted for HAE in the last 3 months and with a medical file.

For the caregiver population:

1. A person identified by the patient as part of their support group and who provides support with the management of the patients HAE (including family members, friends, spouse, etc.)

Exclusion Criteria:

For the patient population:

1. Opposes to participating in the study.
2. Patients is under guardianship or deprived of their liberty.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — All patients, irrespective of their gender are eligible for the study.
Study Population: Patients with HAE
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
To describe the burden associated with the on-demand treatment of HAE attacks | The survey will focus on HAE attacks that have occurred within the last 12 months.
  The burden associated with the on-demand treatment of HAE attacks from the patient's and caregiver's perspective, will be described in terms of:
  * The frequency of HAE attacks.
  * The severity of HAE attacks.
  * Disease control.
  * Events that trigger the HAE attacks.
  * Frequency of injections for treating HAE attacks.
  * Delay in injections for treating HAE attacks.
  * Hospitalization for HAE attacks.
  * Impact on quality of life (during HAE attacks).
  * Impact on quality of life (between HAE attacks).
  * Social impact.
  * Financial impact.
  * Burden of the caregivers.

SECONDARY OUTCOMES:
Use of on-demand treatments for HAE attacks | The survey will focus on HAE attacks that have occurred within the last 12 months.
  The survey will collect data to for the following:
  * To estimate the number of patients that delay or do not use injectable on-demand treatments for HAE.
  * To identify the reasons why patients, delay or do not use injectable on-demand treatments for HAE attacks.
  * To study the potential benefits of introducing an oral on-demand treatment for HAE attacks.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

IPD SHARING:
Plan to Share IPD: Yes
Upon reasonable request.